CLINICAL TRIAL: NCT03773211
Title: Phase I Double Blind Placebo Controlled Safety Study of ex Vivo Treatment of Kidneys From Deceased Donors With Renaparin®, Followed by Transplantation to Study Population
Brief Title: Renaparin® in Kidney Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corline Biomedical AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RENAPAIR 01
Record Dates: First submitted 2018-12-10; First posted 2018-12-12 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Delayed Graft Function
MeSH Terms: conditions — Delayed Graft Function

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Renaparin (Experimental): Solution administered once to kidney ex-vivo
  Interventions: Drug: Renaparin
- Placebo (Placebo Comparator): Placebo administered once to kidney ex-vivo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Renaparin — 50 mL added at one occasion ex-vivo to machine perfusion solution to treat kidney at least 3 hours prior to transplantation
  Arms: Renaparin
Drug: Placebo — 50 mL added at one occasion ex-vivo to machine perfusion solution to treat kidney at least 3 hours prior to transplantation
  Arms: Placebo

SUMMARY:
This study evaluates the safety and tolerability of Renaparin in adult patients receiving a deceased donor kidney treated ex-vivo with Renaparin prior to transplantation. Half the patient group will receive a kidney treated with Renaparin, while the other half of the patient group will receive a kidney treated with placebo.

DETAILED DESCRIPTION:
Kidney transplantation is the last resort for end-stage renal disease (ESRD). A key problem after transplantation is Delayed Graft Function (DGF). Short term, DGF will result in patients being put on dialysis in the immediate time-period after transplantation. In the longer perspective DGF is associated with increased risk of graft failure, thus decreasing the efficacy of the kidney transplantation.

Renaparin is a new product under development for the prevention of DGF in association with kidney transplantation. The product binds to the kidney vascular endothelium and its pharmacological effect is based on a local and effective presentation of heparin. Renaparin is administered ex vivo to the kidney by adding it to the preservation solution during Hypothermic Machine Perfusion (HMP) prior to transplantation.

ELIGIBILITY:
Inclusion Criteria:

Organs:

* Kidney must come from a deceased donor above 18 years of age
* The regular protocols for organ donation according to Swedish law can be followed

Patients:

* Male and female patients 18 - 75 years of age.
* Ability to provide written informed consent.
* Mentally stable and able to comply with the procedures of the study protocol
* Patient has been listed for kidney transplantation from a deceased donor at the clinical sites included in this study.
* Negative crossmatch test prior to transplantation and no existence of donor-specific antibodies
* Receiving first or second renal transplantation

Exclusion Criteria:

Organs:

* Organs from donors deceased due to cardiac death.
* Organs which have not been adequately perfused during HMP, as judged by the transplantation surgeon on call.

Patients:

* Use of an investigational drug or other investigational treatment, that could interfere with the outcome of the present trial, in the 30 days' period before Study Day 1
* Increased risk of thrombosis (ex. homozygous APC-resistance) or bleeding (INR>1.5)
* Anticoagulant treatment with Warfarin for indication unrelated to the kidney transplantation
* History of heparin-induced thrombocytopenia (HIT)
* History of or positive for HIV, HBV, or HCV
* History of oncological malignancy within the last five years, except excised squamous or basal cell carcinoma of the skin
* Scheduled to undergo multi-organ transplantation or dual kidney transplantation
* Current drug and/or alcohol abuse
* Known fish allergy
* History or presence of a medical condition or disease or psychiatric condition that in the investigator's assessment would place the patient at an unacceptable risk for study participation
* Lactating or pregnant women or women who intend to become pregnant
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using effective methods of contraception during study treatment. Acceptable birth control methods are those with a failure rate of less than 1% per year when used consistently and correctly. Such methods include (in "Recommendations related to contraception and pregnancy testing in clinical trials", supplied from www.hma.eu/):

  1. Combined (estrogen and progestogen containing hormonal contraception associated with inhibition of ovulation

     * oral
     * intravaginal
     * transdermal
  2. progestogen-only hormonal contraception associated with inhibition of ovulation

     * oral
     * injectable
     * implantable
  3. intrauterine device
  4. intrauterine hormone-releasing system
  5. bilateral tubal occlusion
  6. vasectomized partner
* Patients who the investigator considers not eligible to give informed consent
* Presence of ECG-based evidence of acute myocardial infarction, unstable angina, decompensated heart failure, third degree of heart block or cardiac arrhythmia associated with hemodynamic stability
* Patients with any condition or any circumstance that in the opinion of the investigator would make it unsafe to undergo a kidney transplantation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2020-04-21 (Actual); Study Completion 2020-04-21 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 30 days
  Number and severity grade of Serious Adverse Events and Adverse Events including description of their associated MedDRA terms during the first 30 days after transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Sedigh, MD, Principal Investigator — Section of Transplantation Surgery, Uppsala University Hospital
Locations (3):
- Sweden (3):
  - Transplantationscentrum, Sahlgrenska University Hospital, Gothenburg
  - Department of Transplantation Surgery, Karolinska University Hospital, Huddinge, Stockholm
  - Department of Surgical Sciences, Section of Transplantation Surgery, Uppsala University Hospital, Uppsala